CLINICAL TRIAL: NCT04937764
Title: Interest of Medial Partial Arthrodesis in Degenerative and Inflammatory Damage of Lisfranc Tarsometatarsal Joint.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Didier MAINARD, Professor, Central Hospital, Nancy, France
Other Study IDs: 2021PI033
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Arthritis Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Population who underwent a surgical arthrodesis procedure for arthritic or inflammatory involvement of the Lisfranc tarsometatarsal joint

SUMMARY:
Research Hypothesis: Lisfranc tarsometatarsal joint arthrodesis is a reliable surgical procedure, allowing the restoration of satisfactory function and a painless foot with an acceptable complication rate.

Objective of the study: To analyze the clinical and radiographic results in the medium term of arthrodesis of the Lisfranc tarsometatarsal joint in cases of primary osteoarthritis, post-traumatic osteoarthritis or in cases of inflammatory pathology.

DETAILED DESCRIPTION:
Data collection by return to the patient record:

* Clinical score
* Analysis of imagery (X-rays, CT scan, )

The patients included were those who had undergone arthrodesis of the medial Lisfranc joint

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent Lisfranc arthrodesis for primary post-traumatic osteoarthritis or inflammatory disease between January 2008 and December 2020 in
* Age > 18 ans

Exclusion Criteria:

* Follow-up < 6 months
* Lost to follow-up
* lack of data in the patient record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent Lisfranc arthrodesis for primary post-traumatic osteoarthritis or inflammatory disease between January 2008 and December 2020 in the department of orthopeadic surgery of the CHU NANCY
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-04-08 (Actual); Primary Completion 2009-01-27 (Actual); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement of the AOFAS score of the midfoot | 1 year post surgery
  AOFAS Score

CONTACTS AND LOCATIONS:
Overall Officials: Didier Mainard, Pr, Study Director — CHU NANCY
Locations (1):
- CHRU NANCY, Central Hospital, Nancy, Meurthe Et Moselle, France

IPD SHARING:
Plan to Share IPD: No
No sharing data